CLINICAL TRIAL: NCT03632564
Title: Modulation of Brain Blood Flow Using Dichoptic Visual and Auditory Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Visior Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SMC-5167-18
Record Dates: First submitted 2018-08-11; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cerebral Arterial Diseases
MeSH Terms: conditions — Cerebral Arterial Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stimulation Arm (Experimental): REVIVIEW dichoptic audio-visual stimulation
  Interventions: Device: REVIVIEW dichoptic audio-visual stimulation

INTERVENTIONS:
Device: REVIVIEW dichoptic audio-visual stimulation — REVIVIEW dichoptic audio-visual stimulation using video goggles

SUMMARY:
Modulation of brain blood flow using dichoptic Visual and Auditory stimulation using REVIVIEW system will be evaluated.

DETAILED DESCRIPTION:
The participant will undergo baseline MRI to measure blood flow in the brain for comparison later on. After baseline MRI, the participant will observe stimulation using the REVIVIEW system for 20 minutes. The content the participants will see is a nature documentary, after which the participant will undergo additional MRI imaging to assess the change in blood flow in the brain.

ELIGIBILITY:
Inclusion Criteria:

- healthy subjects

Exclusion Criteria:

* History of brain diseases
* Glasses
* Diagnosed with Diabetes
* Diagnosed with Degenerative brain diseases
* Inability to undergo MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in blood flow in the brain in respond to the stimulation | 1 hour
  Evaluate the change in blood flow in different parts of the brain, compared with baseline, after the cessation of stimulation, after 30 minutes and after 60 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided